CLINICAL TRIAL: NCT04689477
Title: Non-invasive Characterization of Systemic Microvascular Reactivity by Near-infrared Diffuse Optical Spectroscopy in COVID-19 Patients
Acronym: HEMOCOVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Institut de Ciències Fotòniques (ICFO) (Unknown); Centre de Recerca Matemàtica (Unknown); Institute of Physics University of Campinas (Unknown)
Responsible Party: Principal Investigator, Jaume Mesquida, MD, PhD, Corporacion Parc Tauli
Other Study IDs: 2020/579
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Endothelial Function
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- COVID-19: Hospitalized patients diagnosed with COVID-19, presenting with arterial hypoxemia.
  Interventions: Device: Vascular occlusion test
- Control: Healthy subjects
  Interventions: Device: Vascular occlusion test
- Non-COVID critically ill patients: Non-COVID critically ill patients admitted to the ICU.
  Interventions: Device: Vascular occlusion test

INTERVENTIONS:
Device: Vascular occlusion test — The ischemic challenge will consist in a standardized Vascular Occlusion Test (VOT), as previously described in the literature. Briefly, a blood pressure cuff will be placed proximal to the forearm, and rapidly inflated at 40 mmHg above systolic pressure, and kept inflated during three minutes. Then the cuff will be rapidly deflated. The resulting deoxygenation (DeO2) and reoxygenation (ReO2) slopes will be reported as change in O2 saturation over time.

SUMMARY:
The purpose of this study is to characterize microvascular reactivity on the forearm muscle using non-invasive near-infrared spectroscopy in critically ill COVID-19 patients, and to correlate its alterations with 28-day mortality in ICU COVID-19 patients.

DETAILED DESCRIPTION:
After giving consent to participate in the study, the subjects included in the study will undergo a 15-minute measurement of tissue oxygen saturation (StO2) measured non-invasively on the forearm by means of near-infrared spectroscopy (NIRS). Once a baseline stable StO2 value is obtained, a provocative test, consisting of a transient vascular occlusion, will be performed. The test will allow the obtention of a local metabolic rate, and a StO2 recovery rate after the ischemic stimulus. This StO2 recovery rate will be considered as a reflection of the endothelial health of the patient.

Patients will be studied as soon as possible after admission to the ICU, and followed-up until ICU discharge or death.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of SARS-CoV2 infection
* Arterial hypoxemia and bilateral alveolar infiltrates, not explained by cardiac dysfunction or fluid overload.

Exclusion Criteria:

* Severe peripheral vasculopathy
* Raynaud's syndrome
* Skin lesions or trauma in upper limbs interfering the placement of NIRS probe and/or the occlusion tourniquet
* Deep venous thrombosis in the upper limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critical COVID-19 patients with respiratory impairment admitted to the Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 612 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  Mortality at 28 days of patients admitted to the ICU as results of respiratory failure secondary to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Mesquida, MD, PhD, Principal Investigator — Corporacion Parc Tauli
Locations (8):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States
- Brazil (2):
  - Hospital de Clinicas da UNICAMP, Campinas, São Paulo
  - Hospital Das Clínicas University of Sao Paulo Medical School, São Paulo
- Hospital General de México, México, Mexico
- Spain (4):
  - Institut d'Investigació i Innovació Parc Taulí, Sabadell, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Parc Salut Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona

REFERENCES:
- [Result] Mesquida J, Caballer A, Cortese L, Vila C, Karadeniz U, Pagliazzi M, Zanoletti M, Pacheco AP, Castro P, Garcia-de-Acilu M, Mesquita RC, Busch DR, Durduran T; HEMOCOVID-19 Consortium. Peripheral microcirculatory alterations are associated with the severity of acute respiratory distress syndrome in COVID-19 patients admitted to intermediate respiratory and intensive care units. Crit Care. 2021 Nov 8;25(1):381. doi: 10.1186/s13054-021-03803-2. PMID 34749792
- See also: Related Info — http://hemocovid19-project.org